CLINICAL TRIAL: NCT05270122
Title: ThrombX Retriever for Acute Ischemic Stroke Trial
Acronym: TRAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ThrombX Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T0268
Record Dates: First submitted 2022-02-17; First posted 2022-03-08 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ThrombX Retriever (Experimental): Access to the involved vasculature and preform mechanical thrombectomy using the ThrombX Retriever.
  Interventions: Device: Mechanical thrombectomy with ThrombX Retriever

INTERVENTIONS:
Device: Mechanical thrombectomy with ThrombX Retriever — Revascularization
  Other Names: Mechanical Thrombectomy

SUMMARY:
This trial is designed to assess the safety and effectiveness of the ThrombX Retriever.

DETAILED DESCRIPTION:
This trial is a clinical evaluation is to assess the safety and effectiveness of the ThrombX Retriever in the revascularization of the site of primary occlusion in patients presenting with acute ischemic stroke secondary to intracranial, large vessel, occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

* Acute anterior circulation ischemic stroke
* Pre-stroke Modified Rankin Score ≤ 1
* NIHSS ≥ 6 and < 25 immediately prior to enrollment
* ASPECT score ≥6 with CT scanning or core infarct volume <50 mL on magnetic MRI or CT based perfusion imaging
* Occlusion of IC or the middle cerebral artery M1 or M2 division
* Subject can be treated within eight-hours of onset of stroke symptoms

Exclusion Criteria:

* Pregnant or lactating at time of admission
* Known serious sensitivity to radiographic contrast agents
* Known sensitivity to nickel, titanium metals, or their alloys
* Current participation in another investigation drug or device treatment study
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency prothrombin time lab results to be available prior to enrollment)
* Renal failure
* Baseline blood glucose of <50mg/dL (2.78 mmol/L) or >400mg/dL (22.20 mmol/L)
* Baseline platelet count < 50,000/uL
* Severe, sustained hypertension
* Presumed septic embolus, suspicion of bacterial endocarditis
* Subject has a contraindication to an angiogram
* Life expectancy <6 months
* Comorbid disease or condition that would confound assessments
* Known history of arterial tortuosity, preexisting stent, and/or other arterial disease
* Tandem lesions, occlusion requiring angioplasty and/or stent placement or evidence of carotid dissection
* Site of occlusion is heavily calcified
* Imaging or clinical evidence of bilateral strokes or concomitant posterior circulation stroke
* CT or MRI evidence of hemorrhage or evidence of mass effect or intra-cranial tumor
* Imaging evidence suggests subject is not appropriate for mechanical thrombectomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Successful reperfusion of the occluded target vessel with up to 3 passes of the ThrombX Retriever | Up to the end of theprocedure
  Defined by a mTICI score >2b
Safety Endpoint | 24 hours
  Symptomatic intracerebral hemorrhage (sICH) confirmed on imaging and other Serious Adverse Device Effects (SADE) within 24 hours post procedure. The sICH is defined as the presence of extravascular blood in the cranium associated with an increase in the NIHSS score of ≥ 4 points or death.

SECONDARY OUTCOMES:
Functional independence defined by modified Rankin Scale (mRS) | 90 Days
  modified Ranking Scale is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms to death.

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Jayaraman, MD, Principal Investigator — Rhode Island Hospital; Raul Nogueira, MD, MD, Principal Investigator — University of Pittsburgh Medical Center

IPD SHARING:
Plan to Share IPD: No